CLINICAL TRIAL: NCT06955416
Title: A Multicenter, Randomized, Double-blind Study of the Safety and Efficacy of REAMBERIN®, 1.5% Solution for Infusions, in Addition to Standard Rehydration Therapy in Patients With Diabetic Ketoacidosis
Brief Title: REAMBERIN® 1.5% in Rehydration Therapy of Diabetic Ketoacidosis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RMB-II-III-DKA-2024
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Ketoacidosis
MeSH Terms: conditions — Diabetic Ketoacidosis | interventions — Reamberin

STUDY DESIGN:
Intervention Model Description: A multicenter, prospective, two-stage, comparative, randomized, double-blind, parallel-group study with an adaptive design.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reamberin (Experimental): Infusion of study drug REAMBERIN® for 2 days or until resolution of diabetic ketoacidosis (DKA), whichever occurs first
  Interventions: Drug: Reamberin
- Placebo (Placebo Comparator): Infusion of 0,9% normal saline at the same volume for 2 days or until resolution of diabetic ketoacidosis (DKA), whichever occurs first
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Reamberin — Infusion of study drug REAMBERIN®, solution for infusion 1.5%, in a volume of 750-1500 ml per day (in accordance with the optimal dose established in stage 1), for 2 days or until resolution of DKA, whatever occurs earlier.
  Arms: Reamberin
Drug: Placebo — Infusion of 0,9% normal saline in a volume of 750-1500 ml per day (in accordance with the optimal dose established in stage 1), for 2 days or until resolution of DKA, whatever occurs earlier.
  Arms: Placebo

SUMMARY:
A number of scientific papers have been published on the efficacy and safety of adding REAMBERIN® (meglumin sodium succinate), a 1.5% infusion solution, to standard therapy for patients with diabetic ketoacidosis (DKA), which showed that the addition of the medication to DKA therapy at a dose of 10 ml/kg/day or an average of 800.68±151.59 ml on the first day of infusion, leads to a more rapid and successful resolution of DKA, achieving a state of compensation, a more rapid transfer of the patient from the intensive care unit (ICU) and discharge from the hospital.

A combined, two-stage, multicenter, randomized, double-blind, phase II/III study with an adaptive design is planned. Stage 1 (phase II) will be a sequential evaluation of 2 doses of the study medication (750 ml and 1500 ml) versus placebo. At the 2nd stage of the study (phase III), additional recruitment of patients will be carried out in two groups in a 1:1 ratio to the experimental group or placebo group, to receive the optimal dose in accordance with the result obtained at stage 1.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Male and female patients aged 18-75 years, inclusive.
* Confirmed diagnosis of type 1 or type 2 diabetes mellitus
* Established clinical diagnosis of DKA at the time of admission
* Plasma glucose > 13.9 mmol / l
* Metabolic acidosis (venous blood pH < 7.25)
* Serum bicarbonate < 18 mmol / l
* Ketonuria ≥ ++
* Possibility of randomizing the patient within 2 hours from admission to the hospital.

Exclusion Criteria:

* Known hypersensitivity to any component of the study drug/standard therapy p
* Blood pH ≤ 6.9 or standard bicarbonate level <5 mmol/l
* Previous use of other solutions containing reserve alkalinity carriers (acetate, lactate, malate, fumarate, etc).
* Conditions requiring emergency surgical intervention
* Abdominal surgeries in the last 14 days
* Traumatic brain injury accompanied by cerebral edema.
* Chronic treatment with steroids, atypical antipsychotics, cancer chemotherapy.
* Acute kidney injury
* Chronic kidney disease stage C5
* Liver injury (increase in alanine aminotransferase (ALT), aspartate aminotransferase (AST) levels by more than 5 times the established reference values).
* Acute pancreatitis
* Sepsis
* Severe multiple or combined trauma
* History of malignancy
* Clinically significant cardiovascular diseases (acute coronary syndrome; acute cerebrovascular accident (CVA) or transient ischemic attack (TIA); chronic heart failure class III - IV according to the NYHA classification; severe uncontrolled arrhythmia).
* Body mass index >=40.0
* Alcohol abuse, drug use, drug use.
* Other specific types of diabetes mellitus.
* Previously diagnosed mental illness
* Participation in another clinical trial or the use of drugs/dietary supplements containing succinic acid less than 30 days before inclusion in this study.
* Pregnancy or breastfeeding.
* SARS-CoV-2 infection
* Low systolic blood pressure (BP) (≤70 mmHg) upon admission to hospital or at the time of inclusion in the study.
* Contraindications to the infusion of REAMBERIN of 0.9% sodium chloride solution.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time from initiation of therapy to resolution of diabetic ketoacidosis (DKA) | 48 hours
  Time from the start of therapy with the study drug/placebo as part of standard therapy until resolution of DKA, hours.
  Criteria for resolution of DKA:
  plasma glucose level <11 mmol/l and at least two of the three acid-base balance indicators: bicarbonate ≥ 18 mmol/l, venous pH ≥ 7.3, anion gap ≤ 12 mmol/l.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Kharitonova, MD, PhD, Study Director — STPF "POLYSAN"
Locations (3):
- Russia (3):
  - State Budgetary Institution of Healthcare of the Arkhangelsk Region "First City Clinical Hospital named after E.E. Volosevich", Arkhangelsk
  - Regional budgetary healthcare institution "Ivanovo regional clinical hospital", Ivanovo
  - Kuzbass Clinical Hospital of Emergency Medical Care named after M.A. Podgorbunsky, Kemerovo

IPD SHARING:
Plan to Share IPD: No